CLINICAL TRIAL: NCT04747743
Title: Assessment of Dentist Pharmacist Communication About Usage of Skeletal Muscle Relaxants Survey Among Egyptian Dental Practitioners
Brief Title: Usage of Skeletal Muscle Relaxants Survey Among Egyptian Dental Practitioners
Status: Completed | Type: Observational
Sponsor: Future University in Egypt (Other)
Collaborators: Ain Shams University (Other); British University In Egypt (Other); Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Mohamed Salah ElDin Diab ELBohy, Associate professor, Future University in Egypt
Other Study IDs: FUE.REC 1/1-2021
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Temporomandibular Joint Disorders; Bruxism
MeSH Terms: conditions — Temporomandibular Joint Disorders; Bruxism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Egyptian dental practitioners: 170 dental practitioners in Egypt (professionals both academic and nonacademic).
  Interventions: Other: a self structured questionnaire

INTERVENTIONS:
Other: a self structured questionnaire — A self structured questionnaire to assess knowledge of skeletal muscle use in dental practice

SUMMARY:
Pharmacists may also logistically serve as ideal health-care destinations to implement and deliver prevention, early intervention, and referral of oral health services to reduce the incidence of potentially preventable oral conditions including tooth decay, gum disease, and oral cancer. Interprofessional teamwork between pharmacist and dentistry may help to encourage pharmacists to take a more active role in promoting oral health. By providing information and assistance for self-care and the use of over the counter (OTC) products for minor problems on oral health, it can provide better patient care in the Malaysian health-care system

DETAILED DESCRIPTION:
Skeletal muscle relaxants (SMR) are a diverse group of medications that are not chemically related like other drug classes and work through a variety of mechanisms. The term "muscle relaxant" is used to refer to two major therapeutic groups: neuromuscular blockers and spasmolytic. Some of them are working mainly through the central nervous system; they have many adverse effects such as sedation and dizziness that may limit their use.

Pharmacists may also logistically serve as ideal health-care destinations to implement and deliver prevention, early intervention, and referral of oral health services to reduce the incidence of potentially preventable oral conditions including tooth decay, gum disease, and oral cancer. Interprofessional teamwork between pharmacist and dentistry may help to encourage pharmacists to take a more active role in promoting oral health. By providing information and assistance for self-care and the use of over the counter (OTC) products for minor problems on oral health, it can provide better patient care in the Malaysian health-care system

ELIGIBILITY:
Inclusion Criteria:

* academic dental practitioners in Egypt
* nonacademic dental practitioners in Egypt

Exclusion Criteria:

* Age less than 20 or more than 60
* Non-dental

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: dental practitioners in Egypt (professionals both academic and nonacademic).
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Dental practitioner's knowledge about muscle relaxants indications | 1 month
  Extent of dental practitioner's knowledge about muscle relaxants indications in practice
importance of direct communication between dental practitioners and pharmacists in order to detect the communication barriers and how to overcome those barriers. | 1 month
  To assess and improve the communication between pharmacist- dentist regarding Skeletal muscle relaxant

SECONDARY OUTCOMES:
Dental practitioner's knowledge about muscle relaxants doses | 1 month
  Extent of dental practitioner's knowledge about muscle relaxants different doses in practice
Dental practitioner's knowledge about muscle relaxants side effects | 1 month
  Extent of dental practitioner's knowledge about muscle relaxants possible side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Future University in egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided